CLINICAL TRIAL: NCT01595802
Title: A Non-Randomized, Non-Significant Risk Study Comparing the Nautilus NeuroWaveTM System to Transcranial Doppler as an Aid to Diagnosing Vasospasm
Brief Title: Non-Significant Risk Study Comparing the Nautilus NeuroWaveTM to Transcranial Doppler as an Aid to Diagnosing Vasospasm
Status: Completed | Type: Observational
Sponsor: Jan Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DC1B-01
Record Dates: First submitted 2012-02-14; First posted 2012-05-10 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Vasospasm
Keywords: Cerebral vasospasm
MeSH Terms: conditions — Vasospasm, Intracranial | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects without Vasospasm: Transcranial Doppler (TCD) will be used to evaluate if subject has a vasospasm. Intervention with Nautilus NeuroWave recording to obtain baseline status.
  Interventions: Device: Nautilus NeuroWave; Device: Transcranial Doppler (TCD)
- Subjects with Vasospasm: Transcranial Doppler (TCD) will be used to evaluate if subject has a vasospasm. If confirmed by TCD, the degree of vasospasm will also be evaluated and classified as mild, moderate and severe Vasospasm.
  Intervention with Nautilus NeuroWave recording to obtain recordings with mild, moderate and severe Vasospasm.
  Interventions: Device: Nautilus NeuroWave; Device: Transcranial Doppler (TCD)

INTERVENTIONS:
Device: Nautilus NeuroWave — The Nautilus NeuroWave device will be utilized on subjects with sub-arachnoid hemorrhage that undergo TCD measurements to diagnose Vasospasm. A recording will be obtained using the device each time a TCD measurement is made.
  In this intervention, patients are recorded using the Nautilus Neurowave device.
Device: Transcranial Doppler (TCD) — Subjects with sub-arachnoid hemorrhage undergo TCD measurements to diagnose Vasospasm. Patients that were detected to have a vasospasm using TCD will also be classified as having mild, moderate and severe vasospasm.

SUMMARY:
The purpose of the study is to determine the sensitivity, specificity and predictive values of the Jan Medical NeuroWave System in detecting moderate and severe vasospasm in comparison to Trans Cranial Doppler(TCD).

DETAILED DESCRIPTION:
Cerebral vasospasm generally occurs due to a ruptured brain aneurysm, or (very rarely) hemorrhage from another blood vessel abnormality such as an arteriovenous malformation (AVM). The common factor is the abnormal presence of a substantial amount of blood on the outer ("subarachnoid" or "adventitial") surface of the blood vessel. This can particularly affect arteries at the base of the brain, i.e., around the Circle of Willis.

Depending on the severity, this can be seen using conventional angiography. Angiographic spasm tends to be most readily detected at about 5-7 days after the SAH, although it may be detected as early as 3 days after the hemorrhage. It occurs in between half to two-thirds of all aneurysm patients depending on the time at which angiography was carried out. Clinical vasospasm occurs in approximately one-third of all patients suffering aneurysmal SAH.

The essential problem with vasospasm is that it causes an artery to reduce blood flow or completely shut down. As a result, the part of the brain formerly supplied by that artery effectively starves (ischemia) and may die (infarction or stroke). Overall, cerebral vasospasm accounts for approximately 20% of the severe disability and death associated with ruptured aneurysms.

If vasospasm is detected early, a patient can be treated with balloon angioplasty to reopen the vessels or have infusions of a vasodilator administered (typically verapamil or nicardipine). Alternatively, or in concert with that treatment, one can administer intravenous drugs that raise the patient's blood pressure ("pressors") to force more blood through the narrow arteries. Both of these treatments carry risk and therefore should not be administered unless vasospasm is detected. Therefore, in order to prevent this form of brain injury and enhance the likelihood that a patient will do better, one needs to detect vasospasm before it becomes severe enough to injure the brain.

Vasospasm can be detected by the signs observed on physical examination of the patient and by radiological methods such as cerebral angiography, and Trans-Cranial Doppler (TCD) ultrasound. The physical exam is sensitive for vasospasm in patients who are otherwise awake and able to participate in a neurological examination. Many patients with subarachnoid hemorrhage are not keenly aware nor participative to make this clinical exam meaningful. Therefore clinical examination alone lacks sensitivity.

The gold standard method for detecting vasospasm is cerebral angiography. This involves injection of a radiopaque dye into the arterial blood stream of a patient and when the dye reaches the brain X-rays are taken. Although this is the gold-standard for diagnosing vasospasm it carries the risk of arterial injury or even stroke, and the expense is high. In addition the contrast dye used in these studies carries the risk of renal failure. As a result, this technology is generally employed once vasosapasm is suspected from a Trans Cranial Doppler (TCD) study.

TCD is a bedside test that relies on ultrasound waves generated from a probe placed on the skin of the head and/or neck region to detect the flow of blood in a cerebral artery. It is a convenient, safe, and frequently effective method that can be used to rapidly confirm the clinical findings, and is much less invasive than cerebral angiography. It has, however, numerous technical limitations; for example, one can only detect vasospasm in the proximal vessels of the circle of Willis and therefore lacks sensitivity. It is also quite operator dependent and limited to patients with appropriate skull thickness and acoustic windows.

What is needed is a non-invasive, user independent, safe method to detect cerebral vasospasm before it causes brain injury. The technology needs to be simple to use and can be done at the bedside in an ICU environment. Such a tool will likely improve patient outcome by initiating a chain of events that can mitigate vasospasm (cerebral angioplasty or initiation of vasopressor therapy) and will likely shorten the length of stay within the Neuro ICU saving hospitals money.

The Jan Medical NeuroWave is a simple, rapid, non invasive aid to the diagnosis of vasospasm that is not operator dependent nor limited by skull structure. This study will determine the sensitivity, specificity and predictive values of the Jan Medical NeuroWave System in detecting moderate and severe vasospasm in comparison to Trans Cranial Doppler (TCD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older.
* Subjects with subarachnoid hemorrhage who are receiving clinical and diagnostic surveillance for vasospasm.
* Signed informed consent from the patient or the patient's Legally Authorized Representative

Exclusion Criteria:

* Unstable medical illness such that recordings might interfere with medical care.
* Presence of head bandages or brain monitors that might physically interfere with the tested recording device.
* Current hemicraniectomy.
* Subjects who are not candidates for Transcranial Doppler assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Male or female subjects 18 years of age or older.
  2. Subjects with subarachnoid hemorrhage who are receiving clinical and diagnostic surveillance for vasospasm.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity as a diagnostic aid in detecting vasospasm in subarachnoid hemorrhage | 12 months
  Outcome determine Upon completion of study and unmaksing

SECONDARY OUTCOMES:
Location of vasospasm in the caranium | 12 months
  outcome determine upon completion of study and unmasking
Incidence of device related adverse events | 12 months
  outcome determine upon completion of study and unmasking

CONTACTS AND LOCATIONS:
Overall Officials: Wade Smith, M.D, PH.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco (UCSF), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No